CLINICAL TRIAL: NCT02770703
Title: Mesh Position and Outcomes Following Open (Lichtenstein), Endoscopic (TEP) and Laparoscopic (TAPP) Inguinal Hernia Repair Using a MRI Visible Hernia Mesh
Brief Title: Mesh Position and Outcomes Following Inguinal Hernia Repair Using an MRI Visible Hernia Mesh
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: USB is responsible party on behalf of the principal investigator (PI). As PI cannot be tracked (lost to follow-up), the USB as "sponsor" set "overall recruitment status" unless the PI can be identified or tracked.
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC 2016-00085
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Unilateral Simple Inguinal Hernia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Open inguinal hernia repair (Lichtenstein) (Experimental): Open inguinal hernia repair using a DynaMesh visible mesh
  Interventions: Device: DynaMesh visible mesh
- Total extraperitoneal inguinal hernia repair (TEP) (Experimental): Total extraperitoneal inguinal hernia repair using a DynaMesh visible mesh
  Interventions: Device: DynaMesh visible mesh
- Trans abdominal preperitoneal hernia repair (TAPP) (Experimental): Trans abdominal preperitoneal hernia repair using a DynaMesh visible mesh
  Interventions: Device: DynaMesh visible mesh

INTERVENTIONS:
Device: DynaMesh visible mesh — Implantation of a MRI visible mesh

SUMMARY:
Inguinal hernia repair can be considered as one of the most frequent surgeries in general surgery worldwide. Surgical hernia repair procedures can generally be divided into minimally invasive (TEP, TAPP) and open techniques (e.g. Lichtenstein) and are equivalent with some advantages and disadvantages. The posterior wall of the inguinal channel is usually reinforced by a synthetic mesh, while non-mesh based surgeries have been steadily abandoned.

Two of the most frequent complications following hernia surgery are hernia recurrence and chronic groin pain. Latter can occur in up to 10%. Both represent a considerable socio-economic impact. While different surgical hernia procedures and mesh fixation techniques have been evaluated as influential factors, the impact of mesh position and mesh deformation on hernia recurrence and chronic groin pain is unknown. This may be even more important, since endoscopic and laparoscopic hernia surgery procedures (TEP, TAPP) carry the risk of suboptimal mesh positioning, due to the final steps at the end of the surgery, where the mesh position is not under direct visual control.

Until now direct mesh visualization was impossible. A recent development of MRI visible meshes (DynaMesh® visible) provides the opportunity to evaluate mesh position and deformation after hernia surgery. In case of suspicious clinical hernia recurrence or postoperative chronic groin pain the mesh position can now directly be identified with Magnetic Resonance (MR) imaging preventing unnecessary explorative surgery.

In this study the investigators plan to perform MRI scans to assess mesh position and deformation 90 days postoperatively and correlate it with the clinical status and pain score (VAS) of the patient. In order to allow for an optimal comparison of the post-operative mesh position in relation to the operative technique, patients will be randomized to minimally invasive (TEP, TAPP) and open techniques (e.g. Lichtenstein). To the investigators knowledge this is the first study investigating the impact of the three most common surgical hernia procedures on postoperative mesh position and deformation and its correlation to the clinical findings focussing on hernia recurrence and chronic groin pain.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with a primary symptomatic unilateral inguinal hernia.
* Patients eligible to undergo hernia repair either by minimally invasive (TEP, TAPP) or open techniques (e.g. Lichtenstein) as judged by the treating surgeon
* Written informed consent

Exclusion Criteria:

* Previous inguinal hernia repair
* Bilateral inguinal hernia
* Femoral hernia repair
* Repair in local anesthetics,
* Previous abdominal surgery
* Children
* Emergency surgery, e.g. incarcerated hernias
* Contraindication for MRI scans (e.g. Pacemakers and similar implants, cochlea implants, claustrophobia)
* Contraindications to usage of mesh e.g. known hypersensitivity or allergy
* Women who are pregnant or breast feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia
* American Society of Anesthesiologists (ASA) classification higher or equal to 3

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of Mesh Position per MRI | 90 days postoperatively

SECONDARY OUTCOMES:
Evaluation of Mesh Deformation per MRI | 90 days postoperatively
Groin pain using visual analogue scale | 0, 1, 90, 365 days postoperatively
Recurrence of hernia | 0, 1, 90, 365 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mechera, MD, Principal Investigator — University Hospital of Basel, Department of Surgery
Locations (1):
- University Hospital of Basel, Department of Surgery, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No